CLINICAL TRIAL: NCT05092477
Title: Disease Beliefs and Cognition: Effect on Diabetes Management in Older Breast Cancer Survivors
Brief Title: Integrated Intervention for Breast Cancer Survivors With Diabetes
Acronym: BRIDGES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Northwestern University Feinberg School of Medicine (Other); Feinstein Institute for Medical Research (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jenny J Lin, Professor, General Internal Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: GCO 17-00563; R01CA214491 (NIH)
Record Dates: First submitted 2021-10-13; First posted 2021-10-25 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Diabetes; Breast Cancer
Keywords: Breast Cancer; Intervention; Diabetes; Motivational Interviewing; Cognitive Restructuring; Emotional Response Management
MeSH Terms: conditions — Diabetes Mellitus; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Pilot Overview phase and intervention phase
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant, the outcomes assessor, and the Principal Investigator (Jenny J. Lin) are blinded to study randomization and treatment arm for each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Integrated Intervention (Experimental): 4 intervention sessions over 6 months using an educational and counseling intervention developed by the study team.
  Interventions: Behavioral: Integrated Intervention for Breast Cancer Survivors with Diabetes
- Control (Active Comparator): Attention Control group - Supportive counseling for DM management
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Integrated Intervention for Breast Cancer Survivors with Diabetes — All pilot participants will be required to have a SMB target to be included in this study. A SMB target will be chosen by the participant after reviewing their 18mo follow-up responses with the Care Coach. Participants may endorse a maladaptive belief or emotional response; however, this is not required to participate in this intervention. At each follow-up session, the Care Coach will review the participant's SMB goal and progress, address participant's challenges and suggest alternatives, and correct further misinformation on the disease(s). Additionally, the Care Coach will reinforce or introduce techniques that could help overcome barriers to reaching SMB goal and recommend participants to continue improving on the same goal or begin action planning towards a new SMB goal.
  1. Just SMB concern
  2. SMB + maladaptive belief + emotional response
  3. SMB + maladaptive belief
  4. SMB + emotional response
  Arms: Integrated Intervention
Behavioral: Attention Control — Participants in the control arm will receive a brochure to discuss healthy lifestyle behaviors to improve DM management. To control for the potentially confounding effect of personalized attention from the care coach on the relationship between the intervention and outcomes, participants also receive 4 calls to discuss study progress, thoughts and feelings about study/illness/behaviors, remind them about returning their pill bottles, and about scheduling for their upcoming 24mo follow-up study interview.
  Arms: Control

SUMMARY:
The purpose of this research study is to learn how therapy for breast cancer or DCIS/LCIS affects cognitive function and beliefs about cancer/DCIS/LCIS and diabetes (DM). For this portion of the study, the study team will integrate the information collected at previous follow-ups to create educational modules to change disease and medication beliefs and improve DM self-management behaviors (SMB). The educational counseling modules the study team plans to pilot test are rooted in the Common Sense Self-Regulation Model, a theory that posits that health behaviors are influenced by two parallel processes: cognitive (i.e., disease beliefs and expectations) and affective (i.e., emotional responses).

DETAILED DESCRIPTION:
The study team will develop and pilot an educational and counseling intervention to improve SMB among breast cancer survivors with comorbid DM. Development of Counseling Modules to Promote SMB: The study team will use triangulation analysis to integrate, compare, and contrast the quantitative and qualitative data in order to identify modifiable beliefs and emotional reactions that are associated with DM SMB and which could be the target of tailored education and counseling interventions. The study team will develop modules that address survivors' modifiable beliefs, provide coping skills for emotional reactions to illness, and suggest self-management strategies that have been found to be successful among peers. Triangulation analyses will be conducted following the methods outlined by Farmer beginning with sorting findings from qualitative and quantitative interviews, convergence coding and then convergence assessment, completeness assessment, researcher comparison and feedback.

Developing the Counseling and Education Approach: The CSM has been used to develop behavioral interventions for patients with low adherence to chronic disease SMB. It is similar to DiMatteo's evidence-based 3-factor model of strategies (provide correct information, ensure appropriate beliefs, and eliminate tangible barriers) that has been successfully used to improve medication adherence. The study team will develop 3 basic modules addressing determinants of SMB identified in the study team's quantitative and qualitative analyses and that could be integrated into a future comprehensive self-management support intervention: 1) Addressing DM and Breast Cancer Beliefs: The study team will use cognitive restructuring techniques to address misconceptions about breast cancer and DM and medication adherence. For example, some may believe that DM self-management is not important because breast cancer will likely recur and progress quickly. These views can be "reconstructed" by teaching survivors about timeline and consequences of breast cancer vs. DM allowing them to understand the disease timelines relative to each other. Moreover, the study team will clarify the potential impact of poor DM control on breast cancer outcomes. 2) Addressing Emotional Responses: Anxiety and worries will be addressed with normalizing statements (e.g., "Many patients feel that way..." "It is natural to be worried about side-effects..."). For those who report elevated levels of cancer (or DM) worry and distress, the study team will offer relaxation exercises, such as a deep breathing exercise coupled with stress reducing visualizations. 3) Practical Strategies to Instill Routine SMB: Qualitative interviews will elucidate various strategies that survivors have devised to support their SMB. These patient-identified approaches will be collated and explored with participants as potential strategies the participants might employ as well. Particularly for those with cognitive issues, strategies might include using external aids (i.e., texted phone reminders, alarms, pill box organizers, medication schedules, etc.), linking SMB to routine daily tasks, providing family support, etc. The study team will also use strategies to enhance information comprehension and retention by breast cancer survivors with cognitive dysfunction including teach-to-goal, multi-modal communication, and optimized formatting of print materials.

ELIGIBILITY:
Inclusion Criteria:

* An enrolled participant in the main observational study
* Completed 18-month follow-up interview
* Have at least 1 SMB target (Scored less than scored <4.5 on the MARS for DM, and/or <80% on objective adherence at 12-month (DM), and/or scored <7 on SDSCA)
* Must be willing to participate in the pilot intervention

Exclusion Criteria:

- Participant with suspected clinical depression on CESD (scored ≥20)

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
Illness Perceptions Questionnaire (IPQ scores) | At 6 months
  It is a widely used multi-factorial pencil-and-paper questionnaire which assesses the five cognitive illness representations on a five-point Likert scale. The IPQ is an 80-item instrument, total scale from 0-10, with higher score indicating higher perception of effects on illness.

SECONDARY OUTCOMES:
Medication Adherence (MARS scores) | At 6 months
  To assess beliefs about diabetes medication adherence, the MARS, a validated measure, will be administered after the pilot study, at 6 months. MARS is a 10-item self-reported instrument. Total scores range from 0 (low likelihood of medication adherence) to 10 (high likelihood), with higher score indicating higher likelihood of medication adherence.
Summary of Diabetes Self-Care Activities Assessment (SDSCA) | At 6 months
  The SDSCA measure is a brief self-report questionnaire of diabetes self-management that includes items assessing the following aspects of the diabetes regimen: general diet, specific diet, exercise, blood-glucose testing, foot care, and smoking.
  SDSCA is a validated, self-reported measure assessing the number of days the recommended diabetes self-care activities are performed over the past 7 days in the areas of general diet, specific diet, exercise, blood-glucose testing, and foot care. Possible scores range from 0 to 7 days.
International Physical Activity Questionnaire (IPAQ) | At 6 months
  The purpose of the questionnaires is to provide common instruments that can be used to obtain internationally comparable data on health-related physical activity, a validated measure, will be administered at the end of the pilot study, at 6 months. The IPAQ results can be reported in categories (low activity levels, moderate activity levels or high activity levels) or as a continuous variable (MET minutes a week). MET minutes represent the amount of energy expended carrying out physical activity.
Center for Epidemiological Studies-Depression (CES-D) | At 6 months
  The Center for Epidemiological Studies-Depression (CES-D) is a 20-item measure that asks participants to rate how often over the past week they experienced symptoms associated with depression, such as restless sleep, poor appetite, and feeling lonely. The CES-D also provides cutoff scores (e.g., 16 or greater) that aid in identifying individuals at risk for clinical depression. Full score from 0- 20, with higher score indicating more symptomology.
Objective adherence with eCAP | At 7 months
  The eCAP™ ECM has the regular pharmacy bottle look and feel patients are used to. The important difference is that eCap™ records real-time adherence data, tracking each opening with the date and time.
Beliefs about Medicines Questionnaire (BMQ scores) | At 6 months
  To assess beliefs about medications, the BMQ, a validated measure, will be administered after the pilot study, at 6 months. The BMQ has two components: beliefs about overuse (score range from 3-15) and perceived risk of medicines (score range from 5-25), total scale 8-40, higher score indicates stronger beliefs in the concepts of the scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny J. Lin, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (3):
  - Feinberg School of Medicine, Chicago, Illinois
  - Northwell Health, New Hyde Park, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No
This behavioral coaching intervention plans to enroll a small pilot study of 60 participants. The sample size will be small and the data will be mostly qualitative in nature. The data will be release in the aggregate to protect the participants.